CLINICAL TRIAL: NCT00468325
Title: Coronary Computed Tomography for Systematic Triage of Acute Chest Pain Patients to Treatment (CT-STAT)
Acronym: CTSTAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health East (Other)
Responsible Party: Kavitha Chinnaiyan, MD, William Beaumont Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007-016
Record Dates: First submitted 2007-04-30; First posted 2007-05-02 (Estimated); Last update posted 2009-11-16 (Estimated); Status verified 2009-11

CONDITIONS: Coronary Angiography; Chest Pain
Keywords: coronary artery disease; chest pain; emergency room
MeSH Terms: conditions — Chest Pain; Coronary Artery Disease; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multi-slice Computed Tomography (Active Comparator): Patients admitted to the ED with chest pain and/or anginal equivalent symptoms are randomized to a multi-slice computed tomography arm where they will receive a CT scan of their heart.
  Interventions: Procedure: Multi-slice computed tomography
- Standard of Care (Active Comparator): Patients admitted to the ED with chest pain and/or anginal equivalent symptoms are randomized to the Standard of Care arm and receive rest-stress nuclear myocardial perfusion imaging test.
  Interventions: Procedure: Rest-stress Nuclear Myocardial Perfusion Imaging

INTERVENTIONS:
Procedure: Multi-slice computed tomography — Patient receives a CT scan (multi-slice computed tomography) of the heart.
  Other Names: MSCT; CCTA
  Arms: Multi-slice Computed Tomography
Procedure: Rest-stress Nuclear Myocardial Perfusion Imaging — Patient receives the standard of care for emergency room admitting diagnosis of low to intermediate chest pain. A rest-stress nuclear myocardial perfusion imaging test is performed per the standard of care at each institution.
  Other Names: MPI; Nuclear Stress Test
  Arms: Standard of Care
Procedure: Multi-slice Computed Tomography — Patients admitted to the emergency department with low to intermediate chest pain receive a multi-slice computed tomographic test of the heart.
  Other Names: CCTA; MSCT; Ct Scan of the heart
  Arms: Multi-slice Computed Tomography

SUMMARY:
This is a prospective, randomized multicenter trial comparing MSCT to standard of care (SOC) diagnostic treatment in the triage of Emergency Department (ED) low to intermediate risk chest pain patients. Our hypotheses are that compared to SOC treatment, MSCT is equally safe and diagnostically effective, as well as more time and cost efficient.

DETAILED DESCRIPTION:
Computed tomography (CT) or "cat scan" is an x-ray test routinely used for diagnostic purposes. Heart ("Cardiac") CT, using the newest scanners, is an improved way of looking at the coronary arteries, which supply blood to the heart muscle. If these arteries are clogged this may cause chest pain or even a heart attack. The images of the coronary arteries obtained by CT scanners (during a 5-10 minute procedure) have been shown by many studies to be accurate, when compared to the conventional invasive cardiac catheterization procedure. In addition, at least five prior studies done at different hospitals suggest that cardiac CT scans are effective for diagnosing chest pain like yours in patients coming to the emergency room. What is new about this study is that it is being done in multiple hospitals at the same time. This is part of the process that all medical advances must go through to become a part of routine care of patients in hospitals throughout the country.

A standard chest pain workup typically done in the emergency department consists of a physical examination, electrocardiograms (EKGs), and several blood tests. Blood tests typically completed include cardiac enzymes (Troponin, CK & CK-MB), a kidney function test, a pregnancy test if applicable, and possibly a lipid panel, depending on physician preference. For each test, a 3mL vial will be filled with a specimen of blood and processed in the laboratory for result. Also a two-part "rest-stress" nuclear scan is typically performed, which compares blood flow into the heart tissue at rest to blood flow into the heart tissue during exercise or dilation with medications. Based on prior studies, the researchers doing the present study believe that CT scanning of the coronary arteries can provide information that is just as safe and accurate as the rest-stress nuclear scan, and can do so more rapidly at a lower cost.

ELIGIBILITY:
Inclusion Criteria:

* Chest pain or anginal equivalent symptoms suggestive of acute coronary ischemia within the past 12 hours.
* TIMI risk score less than or equal to 4.
* Ability to provide informed consent.
* Age greater than or equal to 25 years.

Exclusion Criteria:

* Attending physician makes clinical decision for immediate invasive evaluation.
* Electrographic evidence of ischemia, including acute Non ST-Elevation Myocardial Infarction (NSTEMI) or ST-Elevation Myocardial Infarction (STEMI), with ST segment elevation or depression equal to or greater than 1mm in two or more contiguous leads, and/or T wave inversion greater than or equal to 2 mm.
* Positive cardiac biomarkers (troponin, CK, and/or CK-MB) compatible with AMI on initial laboratory testing, based on site standard laboratory values.
* Presence of pre-existing CAD, including prior MI, prior angiographic evidence of significant CAD, defined as greater than or equal to 25% stenosis, or history of coronary artery bypass graft (CABG) surgery.
* Renal insufficiency (creatinine greater than 1.5 mg/dL) or renal failure requiring dialysis.
* Atrial fibrillation or other markedly irregular rhythm.
* Psychological unsuitability or extreme claustrophobia.
* Pregnancy or unknown pregnancy status.
* Clinical instability including cardiogenic shock, hypotension (systolic blood pressure <90 mmHg), refractory hypertension (systolic blood pressure >180 mmHg on therapy), sustained ventricular or atrial arrhythmia requiring intravenous medications.
* Known allergy to iodine or iodinated contrast.
* Inability to tolerate beta-blocker medication, including patients with asthma or chronic obstructive pulmonary disease (COPD) requiring maintenance, i.e. use of inhaled bronchodilators or steroids, or patients with complete heart block or second-degree atrioventricular block.
* Iodinated contrast administration or x-ray scan within the past 48 hours.
* Use of any erectile dysfunction medications such as Viagra or Cialis in the last 24 hours.
* Body Mass Index (BMI) greater than or equal to 39 kg/m2. . Use of biguanides within the past 48 hours

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 750 (Actual)
Dates: Start 2007-05; Primary Completion 2008-11 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Diagnostic efficiency from the time to diagnosis and cost of diagosis for the CCTA and the Standard of Care | Time to diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert Raff, MD, Study Director — Corewell Health East; Kavitha Chinnaiyan, MD, Principal Investigator — Corewell Health East
Locations (16):
- United States (16):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Cleveland Clinic Florida, Weston, Florida
  - Faqua Heart Center/Piedmont Hospital, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan
  - William Beaumont-Troy, Troy, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - St. Paul Heart Clinic, Saint Paul, Minnesota
  - Mt Sinai Hospitl, New York, New York
  - Metrohealth Medical Center, Cleveland, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Heart Institute, Houston, Texas
  - MultiCare Health System-Good Samaritan Hospital, Puyallup, Washington
  - Wisconsin Heart & Vascular Center, Wauwatosa, Wisconsin

REFERENCES:
- [Derived] Goldstein JA, Chinnaiyan KM, Abidov A, Achenbach S, Berman DS, Hayes SW, Hoffmann U, Lesser JR, Mikati IA, O'Neil BJ, Shaw LJ, Shen MY, Valeti US, Raff GL; CT-STAT Investigators. The CT-STAT (Coronary Computed Tomographic Angiography for Systematic Triage of Acute Chest Pain Patients to Treatment) trial. J Am Coll Cardiol. 2011 Sep 27;58(14):1414-22. doi: 10.1016/j.jacc.2011.03.068. PMID 21939822